CLINICAL TRIAL: NCT03407924
Title: Effects of Aerobic Exercise and Rehabilitation After Traumatic Brain Injury
Brief Title: Exercise and Rehabilitation After Traumatic Brain Injury
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Neuro Skills (Industry)
Responsible Party: Principal Investigator, Grace S. Griesbach, National Director of Clinical Research, Centre for Neuro Skills
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AER-TBI1
Record Dates: First submitted 2015-07-09; First posted 2018-01-23 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Exercise; Rehabilitation

STUDY DESIGN:
Intervention Model Description: Intervention will consist of aerobic exercise sessions at predetermined heart rate range.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention aerobic exercise (AER) (Experimental): Participants with traumatic brain injury (TBI) that are enrolled in a comprehensive rehabilitation program (R) will be engaged in an aerobic exercise program (AER). These participants will also receive standard rehabilitation which includes exercise within the physical therapy session. Given that the duration of the rehabilitative program is variable the period of AER training will be no less than 4 weeks and will not exceed 30 weeks. Activity levels will be monitored.
  Interventions: Other: Aerobic Exercise (AER); Other: Rehabilitation
- rehabilitation (R) (Active Comparator): Participants with traumatic brain injury that are enrolled in a comprehensive rehabilitation program. These participants will receive standard rehabilitation. Given that the duration of the rehabilitative program is variable the duration of participation will be no less than 4 weeks and will not exceed 30 weeks. Activity levels will be monitored.
  Interventions: Other: Rehabilitation
- control (C) (No Intervention): Healthy volunteers' responsiveness to exercise and activity levels will be determined to detect TBI effects.

INTERVENTIONS:
Other: Aerobic Exercise (AER) — Aerobic exercise will be performed with a treadmill or stationary tandem bike 3 times per week. Each exercise session will take about 30 minutes plus 5 to 10 min of warm-up and cool-down. Participants will wear a safety harness.
  Arms: Intervention aerobic exercise (AER)
Other: Rehabilitation — Rehabilitative program is focused on completion of activities of daily living, initiation, appropriate behavior and community integration for five days per week at the Centre for Neuro Skills.
  Arms: Intervention aerobic exercise (AER); rehabilitation (R)

SUMMARY:
The purpose of this study is to examine the effects of exercise on recovery after traumatic brain injury. Investigators will determine if exercise enhances rehabilitation by increasing substances (proteins) that can facilitate recovery.

DETAILED DESCRIPTION:
Exercise-based therapies can promote recovery of function and are easily implemented in the clinical rehabilitation setting. This study will determine if exercise facilitates recovery by improving markers of neuroplasticity and decreasing neuroinflammatory responses. The investigators will also determine if variations in genes involved in neuroplasticity, memory and inflammation influence the responsiveness to exercise and rehabilitation. Particular genetic polymorphisms involved in neuroplasticity and inflammatory responses will be evaluated. Recovery will be determined by assessing cognitive function, life quality and balance.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of TBI (for R+AER and R groups).
* Fluency in English or Spanish.
* Able to walk with or without a device.

Exclusion Criteria:

* Orthopedic or cardiac conditions that prevent from exercising.
* Current diagnosis of neurological and/or psychiatric diseases.

Unable to be in the Los Angeles CA metropolitan area for the duration of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-06; Primary Completion 2020-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Aerobic Exercise Induced Changes in Inflammatory responses to exercise | 4 to 30 weeks depending on the duration of rehabilitation coverage.
  Selected analytes will be evaluated from serum.
Aerobic Exercise Induced Changes in Cognitive Function | 5 years
  Attention, processing speed, reaction times, memory and nonverbal reasoning are evaluated by CNS Vital Signs. All scores are aggregated to one reported value (Neurocognitive Index). Scoring is by a computer based auto-scored multivariate scoring system developed by the manufacturers.
Aerobic Exercise Induced Changes in Cardio Pulmonary Fitness | 4 to 30 weeks depending on the duration of rehabilitation coverage.
  Ventilatory Threshold (aerobic capacity)
Aerobic Exercise Induced Changes in Neuroplasticity responses to exercise | 4 to 30 weeks depending on the duration of rehabilitation coverage.
  Selected analytes will be evaluated from serum.

SECONDARY OUTCOMES:
Genetic polymorphisms involved in Inflammatory and neuroplasticity responses to aerobic exercise. | 4 to 30 weeks depending on the duration of rehabilitation coverage.
  Genetic material will be obtained.
Aerobic Exercise Induced Changes in Depression Symptoms | 4 to 30 weeks depending on the duration of rehabilitation coverage.
  Beck Depression Inventory

OTHER OUTCOMES:
Verbal Memory | 4 to 30 weeks depending on the duration of rehabilitation coverage.
  California Verbal Learning Test (CVLT II).
Visual Search/Processing Speed | 4 to 30 weeks depending on the duration of rehabilitation coverage.
  Trail Making
Quality of Life | 4 to 30 weeks depending on the duration of rehabilitation coverage.
  Quality of Life in Neurological Disorders (Neuro-QoL)

CONTACTS AND LOCATIONS:
Overall Officials: Grace S Griesbach, PhD, Principal Investigator — Centre for Neuro Skills
Locations (1):
- Centre for Neuro Skills, Encino, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Griesbach GS, Hovda DA, Molteni R, Wu A, Gomez-Pinilla F. Voluntary exercise following traumatic brain injury: brain-derived neurotrophic factor upregulation and recovery of function. Neuroscience. 2004;125(1):129-39. doi: 10.1016/j.neuroscience.2004.01.030. PMID 15051152
- [Background] Hellawell DJ, Taylor RT, Pentland B. Cognitive and psychosocial outcome following moderate or severe traumatic brain injury. Brain Inj. 1999 Jul;13(7):489-504. doi: 10.1080/026990599121403. PMID 10462147
- [Background] Ashman TA, Gordon WA, Cantor JB, Hibbard MR. Neurobehavioral consequences of traumatic brain injury. Mt Sinai J Med. 2006 Nov;73(7):999-1005. PMID 17195886
- [Background] Alsalaheen BA, Mucha A, Morris LO, Whitney SL, Furman JM, Camiolo-Reddy CE, Collins MW, Lovell MR, Sparto PJ. Vestibular rehabilitation for dizziness and balance disorders after concussion. J Neurol Phys Ther. 2010 Jun;34(2):87-93. doi: 10.1097/NPT.0b013e3181dde568. PMID 20588094
- [Background] Chamelian L, Feinstein A. Outcome after mild to moderate traumatic brain injury: the role of dizziness. Arch Phys Med Rehabil. 2004 Oct;85(10):1662-6. doi: 10.1016/j.apmr.2004.02.012. PMID 15468028
- [Background] Agrawal M, Joshi M. Impact of rehabilitation on functional outcome during the first year of moderate and severe traumatic brain injury. Brain Inj. 2014;28(3):292-7. doi: 10.3109/02699052.2013.865266. Epub 2013 Dec 30. PMID 24378157
- [Background] Griesbach GS, Kreber LA, Harrington D, Ashley MJ. Post-acute traumatic brain injury rehabilitation: effects on outcome measures and life care costs. J Neurotrauma. 2015 May 15;32(10):704-11. doi: 10.1089/neu.2014.3754. Epub 2015 Feb 11. PMID 25496475
- [Background] Chandrasekhar SS. The assessment of balance and dizziness in the TBI patient. NeuroRehabilitation. 2013;32(3):445-54. doi: 10.3233/NRE-130867. PMID 23648599
- [Background] Ridgel AL, Vitek JL, Alberts JL. Forced, not voluntary, exercise improves motor function in Parkinson's disease patients. Neurorehabil Neural Repair. 2009 Jul-Aug;23(6):600-8. doi: 10.1177/1545968308328726. Epub 2009 Jan 8. PMID 19131578